CLINICAL TRIAL: NCT06321471
Title: AeviceMD for Pediatric Asthma Management
Acronym: APAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Irina Dralyuk (Other)
Collaborators: Aevice Health Pte. Ltd. (Other)
Responsible Party: Sponsor-Investigator, Irina Dralyuk, Principal Investigator, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002858
Record Dates: First submitted 2024-03-14; First posted 2024-03-20 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Asthma; Asthma in Children; Pediatric Asthma; Chronic Respiratory Disease
Keywords: Wearable Medical Device
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- AeviceMD (Other): This is a single site, single arm, open label medical device (AeviceMD) pilot where only intervention groups will be recruited.
  Interventions: Device: AeviceMD

INTERVENTIONS:
Device: AeviceMD — AeviceMD is a remote patient monitoring system consisting of a wearable stethoscope, silicone patches, a docking station, and a mobile application.

SUMMARY:
A wearable remote patient monitor (AeviceMD) is to be used to monitor the respiratory health of pediatric asthma patients in this pilot study. Patients prescribed with AeviceMD should be able to gain better control over their disease during home management. Physicians should be able to optimize treatment for these patients using objective data collected from and of these patients outside of the clinic. The AeviceMD should also be used as a remote auscultation device for teleconsultations.

DETAILED DESCRIPTION:
Participants are asked to take part in this research study because they have been diagnosed with poorly controlled asthma. As a chronic respiratory disease, management of the disease relies not only on healthcare professionals delivering care at various clinical touch points, but also depends heavily on a participant's own ability to understand, monitor, and manage their conditions when at home. The investigators know that for pediatric patients, like for many other children, self-monitoring is often difficult. This clinical pilot investigates the use of a wearable medical device that can conduct continuous monitoring of vital signs and detect wheezing when worn at home. The continued use of this device (especially during night sleep) gives insight to the course of symptoms, while also providing early warning should a participant's condition worsen. The device can also be used as a digital stethoscope, meaning physicians can examine participants via teleconference and obtain useful data for clinical decision making.

Study participants include: 20 pediatric patients (between 3 to 18 years of age) who have been diagnosed with poorly controlled asthma while presenting at Cedars-Sinai Medical Center Guerin Children's. Participants will be enrolled to use the AeviceMD device during night sleeps.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Aged 3 to 18 as of first recruitment
* Diagnosed with poorly controlled asthma
* Asthma control test score below
* Caregiver able operate a mobile application
* Has access high-speed wireless internet (WiFi) at home
* Able to read English
* Agreement to adhere to medical device use regimen throughout the study duration

Exclusion Criteria:

* Known allergy to silicone, gold, or zinc
* Abnormal skin conditions on chest
* Sleep apnea diagnosis

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effectiveness of implementing home monitoring technology for asthma patients in delivering care to patients and in extension determine, if Aevice Medical Device can improve home management of Asthma for pediatrics patients. | 3 Months
  The study primary objectives are met if enrolled patients achieve better manage of their asthma shown by a reduction in admission rate, improvement in patient satisfaction, and quality of life. For this purpose, the Pediatric Asthma Control and Communication Instrument (PACCI) system will be utilized. This is a 12-item questionnaire resulting in a sum score ranging from 0 (best asthma control) to 19 (worst asthma control). A decrease in the sum score indicates an improvement in asthma control.

SECONDARY OUTCOMES:
To determine if the AeviceMD is effective as a remote auscultation tool for the facilitation of teleconsultations. | 3 Months
  The study's secondary objectives are met if a remote physician was able to conduct auscultation of a patient's lungs and discern between normal and abnormal breath using AeviceMD during teleconsultations. For this purpose the PI will test the sound quality of the AeviceMD in direct comparison to a traditional stethoscope used at baseline and final in-person visits, as well as at the tele visit.

CONTACTS AND LOCATIONS:
Overall Officials: Irina Dralyuk, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No